CLINICAL TRIAL: NCT03493516
Title: Prediction of ARrhythmic Events With Positron Emission Tomography II
Acronym: PAREPET II
Status: Active, not recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, JOHN CANTY, SUNY Distinguished Professor, State University of New York at Buffalo
Other Study IDs: HL-130266; R01HL130266-01 (NIH)
Record Dates: First submitted 2018-03-26; First posted 2018-04-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-02

CONDITIONS: Sudden Cardiac Arrest; Ischemic Cardiomyopathy; Congestive Heart Failure
Keywords: Positron Emission Tomography; Sympathetic Innervation; Sudden Death; Ventricular Fibrillation; LMI-1195; Ischemic Cardiomyopathy; Risk Prediction
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Failure; Death, Sudden; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples will be obtained for protein biomarkers indicating increased risk of arrhythmias including brain natriuretic peptide levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET scan quantifying sympathetic denervation using [18F]-LMI1195 — A cardiac PET scan will be obtained to quantify the percentage of the left ventricle that is denervated and has reduced uptake of the sympathetic nerve tracer [18F]-LMI1195

SUMMARY:
Sudden cardiac death continues to be a major contributor to mortality in patients with ischemic cardiomyopathy. While implantable defibrillators can prevent death from ventricular arrhythmias, our current approach to identify patients at highest risk primarily rests on demonstrating a reduction in left ventricular ejection fraction less than 35%. The purpose of this observational cohort study is to prospectively test whether this can be enhanced by quantifying the amount of sympathetic denervation, left ventricular end-diastolic volume or brain natriuretic peptide levels.

DETAILED DESCRIPTION:
Using current guidelines based primarily on ejection fraction (EF), only one-quarter of patients receiving an implantable cardiac defibrillator (ICD) for the primary prevention of sudden cardiac arrest (SCA) require appropriate ICD therapy within 5 years. The NIH-sponsored PAREPET study (Prediction of ARrhythmic Events with Positron Emission Tomography, ClinicalTrials.gov, NCT01400334) identified four independent risk factors that predict SCA or ICD equivalent in patients with ischemic cardiomyopathy. Using retrospectively defined cut-points, the absence of these risk factors identified 38% of the cohort with a very low risk of SCA (<1% per year). This rate is actually lower than the 1.5-2% annual rate of SCA among patients with coronary artery disease and mild left ventricular (LV) dysfunction, who are not considered candidates for a primary prevention ICD. This proposal will prospectively determine whether these risk factors can form the basis of a clinically applicable approach to identify a subgroup of patients who are candidates for an ICD, but are at low enough risk of SCA to have an ICD safely withheld. Our long-term goal is to develop better approaches to identify patients with coronary artery disease who are most likely to benefit from prevention of SCA with placement of an implantable defibrillator.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease (by cardiac catheterization or definite myocardial infarction)
* ICD implantation for the primary prevention of SCA
* Primary prevention patients with a Biventricular ICD

  * Eligible immediately when this is placed to prevent dysynchrony related to intermittent RV pacing and the native QRS duration is ≤ 130 msec in the absence of pacing.
  * Eligible 6 months after implantation when the native QRS duration prior to implant is >130 msec or there is persistent RV pacing.
* Optimal medical therapy for heart failure.

Exclusion Criteria:

* Plans for coronary revascularization (due to the independent impact on SCA)
* Contraindication for PET (i.e. claustrophobia, pregnancy, physical limitation)
* Tricyclic antidepressant use (inhibits norepinephrine and LMI1195 uptake)
* Comorbidities limiting life expectancy <2yr.
* Age <18 years or inability to provide informed consent
* Primary prevention ICD/BiV recipients who have received an appropriate ICD shock prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adult patients of either sex with ischemic cardiomyopathy who have an ejection fraction ≤ 35% and New York Heart Association Class II or III CHF or an ejection fraction ≤ 30% and Class I CHF who are candidates to place an ICD for the primary prevention of SCA. Subjects already having a primary prevention ICD are eligible if they have not yet received an appropriate ICD shock for ventricular arrhythmias.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2018-04-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sudden Cardiac Arrest Events | Through study completion, an average of 3 years
  The primary end-point will be SCA or ICD equivalent as used in PAREPET. This will consist of ICD therapies for ventricular fibrillation or ventricular tachycardia >240 bpm, and adjudicated arrhythmic death using the modified Hinkle-Thaler criteria.

OTHER OUTCOMES:
All cause cardiac mortality | Through study completion, an average of 3 years
  Adjudicated total cardiac mortality (SCA + non-sudden cardiac death).
All appropriate ICD therapies | Through study completion, an average of 3 years
  Adjudicated appropriate ICD therapies (ICD shock and anti-tachycardia pacing) for ventricular arrhythmias. Appropriate ICD therapies will be determined from ICD device interrogation.
Hospitalization for heart failure and myocardial infarction. | Through study completion, an average of 3 years
  Interval hospitalizations for heart failure or myocardial infarction will be assessed via phone follow-up at 3 month intervals. Subjects having either will be invited to return for a repeat PET scan, echocardiogram and serum sampling to assess whether the underlying substrate for arrhythmogenesis has changed.

CONTACTS AND LOCATIONS:
Overall Officials: John M Canty, MD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo Clinical and Translational Research Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fallavollita JA, Dare JD, Carter RL, Baldwa S, Canty JM Jr. Denervated Myocardium Is Preferentially Associated With Sudden Cardiac Arrest in Ischemic Cardiomyopathy: A Pilot Competing Risks Analysis of Cause-Specific Mortality. Circ Cardiovasc Imaging. 2017 Aug;10(8):e006446. doi: 10.1161/CIRCIMAGING.117.006446. PMID 28794139
- [Background] Malhotra S, Canty JM Jr. Life-Threatening Ventricular Arrhythmias: Current Role of Imaging in Diagnosis and Risk Assessment. J Nucl Cardiol. 2016 Dec;23(6):1322-1334. doi: 10.1007/s12350-015-0392-0. Epub 2016 Jan 15. PMID 26780530
- [Background] Goldberger JJ, Basu A, Boineau R, Buxton AE, Cain ME, Canty JM Jr, Chen PS, Chugh SS, Costantini O, Exner DV, Kadish AH, Lee B, Lloyd-Jones D, Moss AJ, Myerburg RJ, Olgin JE, Passman R, Stevenson WG, Tomaselli GF, Zareba W, Zipes DP, Zoloth L. Risk stratification for sudden cardiac death: a plan for the future. Circulation. 2014 Jan 28;129(4):516-26. doi: 10.1161/CIRCULATIONAHA.113.007149. No abstract available. PMID 24470473
- [Background] Fallavollita JA, Heavey BM, Luisi AJ Jr, Michalek SM, Baldwa S, Mashtare TL Jr, Hutson AD, Dekemp RA, Haka MS, Sajjad M, Cimato TR, Curtis AB, Cain ME, Canty JM Jr. Regional myocardial sympathetic denervation predicts the risk of sudden cardiac arrest in ischemic cardiomyopathy. J Am Coll Cardiol. 2014 Jan 21;63(2):141-9. doi: 10.1016/j.jacc.2013.07.096. Epub 2013 Sep 25. PMID 24076296

DOCUMENTS (1):
  • Informed Consent Form (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT03493516/ICF_000.pdf